CLINICAL TRIAL: NCT06975787
Title: A Dose Escalation Study Investigating Bispecific Antibody Therapy in Patients With Lupus Nephritis
Brief Title: Dose Escalation Study With Bispecific Antibodies in Adult Patients With Lupus Nephritis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: R5459-1979-LN-2459; 2024-518288-37-00 (EU CTIS Number)
Record Dates: First submitted 2025-05-08; First posted 2025-05-16 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Lupus Nephritis (LN)
Keywords: Bispecific Antibodies (bsAb); Double-stranded DNA (dsDNA); LN class III or IV; Systemic Lupus Erythematosus (SLE)
MeSH Terms: conditions — Lupus Nephritis; Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental Arm 1: Vonsetamig (Experimental)
  Interventions: Drug: Vonsetamig
- Experimental Arm 2: Odronextamab (Experimental)
  Interventions: Drug: Odronextamab

INTERVENTIONS:
Drug: Vonsetamig — Administered as per the protocol
  Other Names: REGN5459
  Arms: Experimental Arm 1: Vonsetamig
Drug: Odronextamab — Administered as per the protocol
  Other Names: REGN1979
  Arms: Experimental Arm 2: Odronextamab

SUMMARY:
This study is researching a particular group of experimental drugs administered for a short period in the treatment of patients with Lupus Nephritis (LN).

The main aim of the current study is to see how safe and tolerable the study drugs are in a long-term follow-up.

This is a main study, called an umbrella study, which includes several independent smaller sub-studies. Each of these smaller main sub-studies tests different drugs at the same time, all aimed at treating LN.

The study is looking at several other research questions, including:

* What side effects may happen from taking the study drug
* How much study drug is in the blood at different times
* Whether the body makes antibodies against the study drug (which could make the drug less effective or could lead to side effects)

ELIGIBILITY:
Key General Inclusion Criteria:

1. Diagnosis of Systemic Lupus Erythematosus (SLE) and LN, as described in the protocol
2. Participant must have refractory or relapsed disease, as described in the protocol

Key General Exclusion Criteria:

1. History of or active severe or unstable lupus-associated neuropsychiatric disease that is likely to require acute or emergent medical treatment or hospitalization
2. Active overlap syndrome with mixed connective tissue disease or systemic sclerosis within 12 months prior to screening or during screening
3. Catastrophic or severe antiphospholipid syndrome within 12 months prior to screening or during screening

NOTE: Other protocol defined inclusion/exclusion criteria apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-12-22 (Actual); Primary Completion 2028-07-23 (Estimated); Study Completion 2028-07-23 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Dose Limiting Toxicities (DLT) | Up to 56 days
Occurrence of Treatment Emergent Adverse Events (TEAEs) | Through week 76
Severity of TEAEs | Through week 76

SECONDARY OUTCOMES:
Proportion of participants receiving a corticosteroid dose of 0 mg per day | At 6 months
Cumulative total exposure to corticosteroids | At 76 weeks
Absolute values of urine Protein-Creatinine Ratio (uPCR) | Through week 76
Percent change from baseline of uPCR | Through week 76
Absolute values of estimated Glomerular Filtration Rate (eGFR) serum creatinine | Through week 76
Percent change from baseline of eGFR serum creatinine | Through week 76
Absolute values of blood B-cell counts and other immune cell populations | Through week 76
  T cells and Natural Killer (NK) cells
Change from baseline of blood B-cell counts and other immune cell populations | Through week 76
  T cells and NK cells
Absolute values of double-stranded DNA (dsDNA) antibodies | Through week 76
Percent change from baseline of dsDNA antibodies | Through week 76
Absolute values of anti-Smith antibodies | Through week 76
Percent change from baseline of anti-Smith antibodies | Through week 76
Absolute values of anti-C1q antibodies | Through week 76
Percent change from baseline of anti-C1q antibodies | Through week 76
Absolute values of other autoantibodies | Through week 76
  anti-nucleosome
Percent change from baseline of other autoantibodies | Through week 76
  anti-nucleosome
Absolute values of Complement Factor C3 (C3) circulating factors | Through week 76
Percent change from baseline of C3 circulating factors | Through week 76
Absolute values of Complement Factor C4 (C4) circulating factors | Through week 76
Percent change from baseline of C4 circulating factors | Through week 76
Absolute values of serum levels of Immunoglobulin A (IgA) | Through week 76
Percent change from baseline of serum levels of IgA | Through week 76
Absolute values of serum levels of Immunoglobulin G (IgG) | Through week 76
Percent change from baseline of serum levels of IgG | Through week 76
Concentrations of vonsetamig in serum over time | Through week 76
Concentrations of odronextamab in serum over time | Through week 76
Incidence of Anti-Drug Antibodies (ADAs) to vonsetamig | Through week 76
Incidence of ADAs to odronextamab | Through week 76
Titer of ADAs to vonsetamig | Through week 76
Titer of ADAs to odronextamab | Through week 76

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (4):
- University Medical Center of the Johannes Gutenberg-University Mainz, Mainz, Germany
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/